CLINICAL TRIAL: NCT03047759
Title: Comparison of Two Interdental Cleaners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All Sum Research Center Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-WP-2
Record Dates: First submitted 2016-08-17; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-08

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Intervention A (Active Comparator): water flosser
  Interventions: Device: water flosser
- Intervention B (Active Comparator): air floss
  Interventions: Device: air floss

INTERVENTIONS:
Device: water flosser — Powered
  Arms: Intervention A
Device: air floss — Powered
  Arms: Intervention B

SUMMARY:
Comparison of Two interdental cleaning devices on plaque removal, gingivitis and bleeding.

DETAILED DESCRIPTION:
This study measured plaque accumulation, bleeding on probing and gingivitis using the Rustogi Modification of the Navy Plaque Index, BOP and Modified Gingival Index at baseline, 2-weeks and 4-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* Non smoker
* Available for 4-weeks
* Able to provide written informed consent.
* Minimum of 20 natural teeth.
* Minimum requirement for plaque, gingivitis and bleeding.

Exclusion Criteria:

* Medical condition
* No antibiotics within 6 months of study start
* Not on any medication (impact oral health).

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-19 (Actual)

PRIMARY OUTCOMES:
Bleeding upon probing | 4 weeks
  Bleeding upon probing

SECONDARY OUTCOMES:
Gingivitis | 4 weeks
  Modified Gingival \index
Plaque | 4 weeks
  Rustogi Modification of the Navy Plaque Index

IPD SHARING:
Plan to Share IPD: No